CLINICAL TRIAL: NCT00374348
Title: "Aripiprazole in the Treatment of Patients With Schizophrenia and Symptoms of Obsessive Compulsive Disorder (OCD)".
Brief Title: Aripiprazole in the Treatment of Patients With Schizophrenia and Symptoms of Obsessive Compulsive Disorder (OCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jamaica Hospital Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Department of Psychiatry, Jamaica Hospital Medical Center (Unknown); Research Division (Ambiguous)
Responsible Party: Isak Isakov, MD, Department of Psychiatry Research Division
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JH-PSY-Aripiprazole/Schiz/OCD
Record Dates: First submitted 2006-09-07; First posted 2006-09-11 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2009-01

CONDITIONS: Schizophrenia OCD; Obsessive Compulsive Disorder
Keywords: Schizophrenia with OCD; Schizophrenia with-comorbid symptoms of Obsessive Compulsive Disorder(OCD)
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Abilify, 5mg; 10mg; 15mg; 20mg; 30mg
  Other Names: Abilify

SUMMARY:
To evaluate the effectiveness of flexible doses (15-30mg) of Aripiprazole in the treatment of patients with schizophrenia and co-morbid symptoms of OCD in the outpatient setting. The overall effectiveness of Aripiprazole will be evaluated by use of the Brief Psychiatric Rating Scale(BPRS), Yale-Brown OCD scale and Clinical Global Impression-Improvement(CGI-I) scale.

DETAILED DESCRIPTION:
Symptoms of OCD is a rather common co-morbid condition in patients with Schizophrenia. Some studies suggest that obsessive-compulsive symptoms may be present in 7.8-46% of schizophrenic patients and who seem to be poorly responsive to drug therapy. The serotonergic medications in combination with cognitive-behavioral therapy stil remain the preferred treatment for OCD symptoms. There are controversial data regarding effect of neuroleptics on symptoms of OCD. It was noted that the use of Risperdone, Quatiapine and Clozapine might aggravate OCD symptoms. Serotonin antagonism of these neuroleptics is believed to exacerbate obsessive-compulsive symptoms in schizophrenia. On the other hand, Pourovsky M. at(2000) reported three cases of Schizophrenia with symptoms of OCD successfully treated with Olanzapine.One of our patients with Schizophrenia and co-morbid symptoms of OCD who was unsuccessfully treated with various neuroleptics in combination with anti-obsessive agents,demonstrated significant improvement in both Schizophrenic and obsessive compulsive symptoms after she was switched to Aripiprazole. This result encouraged us to initiate pilot study of effectiveness of Aripiprazole in the treatment of specific population of schizophrenic patients with symptoms of OCD.

ELIGIBILITY:
Inclusion Criteria:

* Man and Women 18-65 years of age.
* Patients who are capable of giving Informed Consent and fluent in English.
* Patients who have DSM IV -Diagnosis of schizophrenia with co-morbid OCD symptoms and BPRS score averaging from mild to moderate (3-4).
* Patients whose obsessive symptoms are not optimally controlled and require a change of treatment.YBOCS score of more than 16.

Exclusion Criteria:

* Outside the age range of 18-65 years.
* Patients with current evidence(past three months) of substance abuse.
* Women of child bearing age who are unwilling to use acceptable methods of contraception.
* Patients who have had recent treatment with long-acting antipsychotic.
* Patients who are suicidal or who have history of recent suicidal attempt.
* History of significant medical condition e.g. seizures, cardiovascular, endocrine,gastrointestinal,renal or respiratory diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The overall effectiveness of Aripiprazole will be evaluated by use of the BPRS, Yale-Brown OCD scale and Clinical Global Impression-Improvement (CGI-I) scale, including efficacy in reduction of psychosis and obsessions.Improvements in YBOCS and BPRS scor | weekly

SECONDARY OUTCOMES:
Physical Examination, Psychiatric evaluation with YBOCS, BPRS and CGI scales, EPS scale, routine hematology and chemistry tests, urinalysis,urine drug screening,urine pregnancy test, ECG recording | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Isak Isakov, M.D., Principal Investigator — Jamaica Hospital Medical Center
Locations (1):
- Jamaica Hospital Medical Center Department of Psychiatry, Jamaica, New York, United States